CLINICAL TRIAL: NCT01188226
Title: Evaluation of Wear Characteristics of Nano-Hybrid Denture Teeth
Brief Title: Wear Characteristics of Denture Teeth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties and drop outs
Sponsor: University of California, Los Angeles (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Neal Garrett, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101960
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Dentures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nano Hybrid Composite Denture teeth (Experimental): Denture teeth are made of nano hybrid composite material
  Interventions: Device: Denture teeth

INTERVENTIONS:
Device: Denture teeth — Denture teeth made of nano hybrid composite material
  Other Names: Ivoclar Vivadent Inc. SR Phonares denture teeth

SUMMARY:
The majority of teeth utilized in the fabrication of conventional complete dentures are made of acrylic resins. These acrylic teeth provide increased bond strength to the denture base and are much easier to adjust for correct denture occlusion compared to teeth made of harder materials, such as porcelain. However, the acrylic teeth will wear faster than the porcelain teeth, leading to alterations in how the teeth contact each other if the denture is not replaced periodically (typically every 5-8 years). With the increase in biting and chewing forces that can be achieved during function with dentures supported by dental implants, the rate of tooth wear may be increased, leading to more frequent need for replacement of the prosthesis. Acrylic teeth made of nano hybrid composite material (NHC) potentially offer greater wear resistance and aesthetic characteristics. The NHC teeth employ a wide range of fillers, including highly cross-linked organic macrofillers, high-density inorganic microfillers and silanized silica based nanofillers. The macrofillers are, to a large part, responsible for the adequate strength and color-stability of the teeth, whereas the microfillers improve the wear resistance. The nanofillers offer fundamentally different optical behaviour from those of larger fillers, improving light reflection without lowering the translucency. This offers additional opportunities in the development of composite teeth, which have to exhibit lifelike aesthetics and translucency. These teeth made of nano-particles and hybrid composites can be made with two different techniques, one where the materials are pressed together and another using an injection technique. The injection method has been found to have better aesthetic results, but resistance to wear in clinical use has not been established.

The purpose of this study is to evaluate the wear characteristics of new resin denture teeth (nano particles - hybrid composite) made by an injection technique. Twenty-four edentulous subjects will be enrolled who have completed implant placement for mandibular implant overdentures opposing a maxillary complete denture or implant overdenture, or patients that have previously received these dentures and are interested in having new dentures. Both maxillary and mandibular dentures will be fabricated using injection molded nano-hybrid composite denture teeth. The wear of denture teeth will be evaluated using stereophotographic recordings at baseline, 6, 12, 18 and 24 months after denture treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being treated at UCLA School of Dentistry clinics with implant-assisted mandibular overdentures and conventional maxillary complete dentures or implant overdentures
* Previously treated at UCLA School of Dentistry clinics with implant-assisted mandibular overdentures and conventional maxillary complete dentures or implant overdentures and desires new dentures
* Have healthy, normal soft and hard oral tissues

Exclusion Criteria:

* Oral and medical conditions which would interfere with follow-up evaluations over a two-year period after denture treatment completion
* Abnormal oral soft or hard tissues that prevents conventional denture fabrication
* Impaired dexterity the prevents proper oral hygiene
* Allergy to denture base materials
* Severe parafunction based on current condition of existing dentures
* Any limitation in mouth opening or closing
* Severe TMD symptoms
* Employees (and their immediate families) of the UCLA School of Dentistry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Garret, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA School of Dentistry, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nano Hybrid Composite Denture Teeth
Started | 10
Completed | 6
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Subjects that signed consent
Arm/Group | Nano Hybrid Composite Denture Teeth
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Location of Posterior Denture Tooth Wear
Description: Clinical evaluation of posterior wear location (right, left, equal).
Time Frame: 6 months after denture completion
Population: For study participants who completed the 6-month follow-up. Upper and lower dentures of each participant assessed and reported separately as Arms for this outcome.
Measure: Number; unit: participants
Groups:
- Upper Denture; Lower Denture: Denture teeth are made of nano hybrid composite material
Arm/Group | Upper Denture | Lower Denture
Number analyzed (Participants) | 8 | 8
participants
  Right side wear | 0 | 0
  Equal wear | 7 | 6
  Left side wear | 1 | 2

2. Primary Outcome: Location of Posterior Denture Tooth Wear
Description: Clinical evaluation of posterior wear location (right, left, equal)
Time Frame: 12 months after denture completion
Population: For study participants who completed the 12-month follow-up. Upper and lower dentures assessed and reported separately as Arms for this outcome.
Measure: Number; unit: participants
Arm/Group | Upper Denture | Lower Denture
Number analyzed (Participants) | 7 | 7
participants
  Right side wear | 0 | 1
  Equal wear | 6 | 5
  Left side wear | 1 | 1

3. Primary Outcome: Location of Posterior Denture Tooth Wear
Description: Clinical evaluation of posterior wear location (right, left, equal)
Time Frame: 18 months after denture completion
Population: For study participants who completed the 18-month follow-up. Upper and lower dentures of each participant assessed and reported separately as Arms for this outcome.One participant had the lower denture refabricated after 12 months and was not included in 18-month lower-denture assessment
Measure: Number; unit: participants
Groups:
- Lower Denture: Participants with lower denture in use 18 months after denture completion. Denture teeth are made of nano hybrid composite material
Arm/Group | Upper Denture | Lower Denture
Number analyzed (Participants) | 4 | 3
participants
  Right side | 0 | 0
  Equal | 3 | 2
  Left side | 1 | 1

4. Primary Outcome: Location of Posterior Denture Tooth Wear
Description: Clinical evaluation of posterior wear location (right, left, equal)
Time Frame: 24 months after denture completion
Population: For study participants who completed the 24-month follow-up. Upper and lower dentures of each participant assessed and reported separately as Arms for this outcome.One participant had the lower denture refabricated after 12 months and was not included in 24-month lower-denture assessment
Measure: Number; unit: participants
Groups:
- Upper Denture: Participants wearing upper denture 24 months after denture completion. Denture teeth are made of nano hybrid composite material.
- Lower Denture: Participants wearing lower denture 24 months after denture completion. Denture teeth are made of nano hybrid composite material.
Arm/Group | Upper Denture | Lower Denture
Number analyzed (Participants) | 6 | 5
participants
  Right side | 0 | 0
  Equal | 5 | 5
  Left side | 1 | 0

5. Secondary Outcome: Denture Teeth Esthetics
Description: Clinical evaluation of color deviation of anterior teeth to shade guide (3 levels: high, little, none)
Time Frame: 6 months after denture completion
Measure: Number; unit: participants
Groups:
- Participants With Nano Hybrid Composite Dentures: Denture teeth are made of nano hybrid composite material
Arm/Group | Participants With Nano Hybrid Composite Dentures
Number analyzed (Participants) | 8
participants
  Deviation: High | 0
  Deviation: Little | 2
  Deviation: None | 6

6. Secondary Outcome: Amount of Denture Teeth Plaque
Description: Clinical evaluation of plaque for anterior teeth and left posterior teeth and right posterior teeth on four-point scale (0= none; 1 = soft debris covering ≤1/3 of tooth surface; 2 = soft debris covering > 1/3 and ≤ ½ of tooth surface; 3 = soft debris covering more than ½ of tooth surface)
Time Frame: 6 months after denture completion
Population: For study participants who completed the 6-month follow-up. Anterior, right-posterior, and left-posterior denture teeth areas of each participant assessed and reported separately as Arms for this outcome.
Measure: Number; unit: participants
Groups:
- Anterior Denture Teeth; Right-posterior Denture Teeth; Left-posterior Denture Teeth: Denture teeth are made of nano hybrid composite material
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 8 | 8 | 8
participants
  0=None | 5 | 5 | 5
  1=Soft debris covering ≤1/3 of surface | 2 | 2 | 2
  2=soft debris covering > 1/3 and ≤ ½ of surface | 1 | 1 | 1
  3=soft debris covering more than ½ of surface | 0 | 0 | 0

7. Secondary Outcome: Denture Teeth Calculus
Description: Clinical evaluation of calculus for anterior teeth and posterior teeth on left and right sides on four-point scale (0= none; 1 = present on ≤ 1/3 of gingival margins; 2 = present on > 1/3 of gingival margins and parts of fissures and/or individual spots around cervical portion of tooth; 3 = covering more than ½ of gingival margins and the complete fissures and/or continuous heavy band of calculus around cervical portion of the tooth)
Time Frame: 6 months after denture completion
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 8 | 8 | 8
participants
  0 | 8 | 8 | 8
  1 | 0 | 0 | 0
  2 | 0 | 0 | 0
  3 | 0 | 0 | 0

8. Secondary Outcome: Denture Teeth Esthetics
Description: Clinical evaluation of color deviation of anterior teeth to shade guide (3 levels, high, little none)
Time Frame: 12 months after denture completion
Population: For study participants who completed the 12-month follow-up.
Measure: Number; unit: participants
Arm/Group | Nano Hybrid Composite Denture Teeth
Number analyzed (Participants) | 7
participants
  Deviation: High | 1
  Deviation: Little | 2
  Deviation: None | 4

9. Secondary Outcome: Denture Teeth Esthetics
Description: Clinical evaluation of color deviation of anterior teeth to shade guide (3 levels: high, little, none)
Time Frame: 18 months after denture completion
Population: For study participants who completed the 18-month follow-up.
Measure: Number; unit: participants
Arm/Group | Nano Hybrid Composite Denture Teeth
Number analyzed (Participants) | 4
participants
  Deviation: High | 0
  Deviation: Little | 1
  Deviation: None | 3

10. Secondary Outcome: Denture Teeth Esthetics
Description: Clinical evaluation of color deviation of anterior teeth to shade guide (3 levels: high, little, none)
Time Frame: 24 months after denture completion
Population: For study participants who completed the 24-month follow-up.
Measure: Number; unit: participants
Arm/Group | Nano Hybrid Composite Denture Teeth
Number analyzed (Participants) | 6
participants
  Deviation: High | 1
  Deviation: Little | 3
  Deviation: None | 2

11. Secondary Outcome: Amount of Denture Teeth Plaque
Description: as for outcome 6
Time Frame: 12 months after denture completion
Population: For study participants who completed the 12-month follow-up. Anterior, right-posterior, and left-posterior denture teeth areas of each participant assessed and reported separately as Arms for this outcome.
Measure: Number; unit: participants
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 7 | 7 | 7
participants
  0= none | 6 | 6 | 5
  1 = soft debris covering ≤1/3 of tooth surface | 1 | 1 | 2
  2 = soft debris covering > 1/3 and ≤ ½ of surface | 0 | 0 | 0
  3 = soft debris covering more than ½ of surface | 0 | 0 | 0

12. Secondary Outcome: Amount of Denture Teeth Plaque
Description: as for outcome 6
Time Frame: 18 months after denture completion
Population: For study participants who completed the 18-month follow-up. Anterior, right-posterior, and left-posterior denture teeth areas of each participant assessed and reported separately as Arms for this outcome.
Measure: Number; unit: participants
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 4 | 4 | 4
participants
  0 = None | 3 | 4 | 4
  1 = soft debris covering ≤1/3 of tooth surface | 1 | 0 | 0
  2 = soft debris covering > 1/3 and ≤ ½ of surface | 0 | 0 | 0
  3 = soft debris covering more than ½ of surface | 0 | 0 | 0

13. Secondary Outcome: Amount of Denture Teeth Plaque
Description: as for outcome 6
Time Frame: 24 months after denture completion
Population: For study participants who completed the 24-month follow-up. Anterior, right-posterior, and left-posterior denture teeth areas of each participant assessed and reported separately as Arms for this outcome.
Measure: Number; unit: participants
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 6 | 6 | 6
participants
  0 = None | 5 | 4 | 4
  1 = soft debris covering ≤1/3 of tooth surface | 0 | 2 | 2
  2 = soft debris covering > 1/3 and ≤ ½ of surface | 1 | 0 | 0
  3 = soft debris covering more than ½ of surface | 0 | 0 | 0

14. Secondary Outcome: Denture Teeth Calculus
Description: as for outcome 7
Time Frame: 12 months after denture completion
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 7 | 7 | 7
participants
  0 | 6 | 6 | 6
  1 | 1 | 1 | 1
  2 | 0 | 0 | 0
  3 | 0 | 0 | 0

15. Secondary Outcome: Denture Teeth Calculus
Description: as for outcome 7
Time Frame: 18 months after denture completion
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 4 | 4 | 4
participants
  0 | 4 | 4 | 4
  1 | 0 | 0 | 0
  2 | 0 | 0 | 0
  3 | 0 | 0 | 0

16. Secondary Outcome: Denture Teeth Calculus
Description: as for outcome 7
Time Frame: 24 months after denture completion
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Anterior Denture Teeth | Right-posterior Denture Teeth | Left-posterior Denture Teeth
Number analyzed (Participants) | 6 | 6 | 6
participants
  0 | 6 | 4 | 4
  1 | 0 | 2 | 2
  2 | 0 | 0 | 0
  3 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Nano Hybrid Composite Denture Teeth
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nano Hybrid Composite Denture Teeth (N=10)
Denture tooth fracture (Gastrointestinal disorders) | 6 (11) — One tooth or multiple teeth fractured and repaired during study
Lower denture break (Gastrointestinal disorders) | 1 (1) — Lower denture broke at midline and was replaced during the study
Tooth debonding (Gastrointestinal disorders) | 1 — Tooth debonding requiring recementation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No